CLINICAL TRIAL: NCT01963039
Title: A Randomised Sham Controlled Trial of Vertebroplasty for Painful Chronic Osteoporotic Vertebral Fractures
Brief Title: A Trial of Vertebroplasty for Painful Chronic Osteoporotic Vertebral Fractures (Vertos V)
Acronym: VERTOSV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elisabeth-TweeSteden Ziekenhuis (Other)
Collaborators: Stryker Medical (Industry); Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EZTilburg2
Record Dates: First submitted 2013-08-28; First posted 2013-10-16 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Osteoporosis; Vertebral Fracture
MeSH Terms: conditions — Osteoporosis; Spinal Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- percutaneous vertebroplasty (Active Comparator): Using fluoroscopic guidance, the practitioner infiltrates the skin and subcutaneous tissues overlying the pedicle of the target vertebra or vertebrae with 1% lidocaine and infiltrates the periosteum of the pedicles with 0.25% bupivacaine (marcaine). For the vertebroplasty procedure, 11-gauge or 13-gauge needles are passed into the central aspect of the target vertebra or vertebrae. Bone cement (PMMA) is prepared on the bench and injected under constant fluoroscopy into the vertebral body. Injection is stopped when the cement reaches to the posterior aspect of the vertebral body or leaks into an extraosseous space, such as the intervertebral disk or an epidural or paravertebral vein.
  Interventions: Device: percutaneous vertebroplasty
- Sham procedure (Sham Comparator): Using fluoroscopic guidance, the practitioner infiltrates the skin and subcutaneous tissues overlying the pedicle of the target vertebra or vertebrae with 1% lidocaine and infiltrates the periosteum of the pedicles with 0.25% bupivacaine (marcaine). During the sham intervention, verbal and physical cues, such as pressure on the patient's back, are given, and the bone cement(PMMA) is prepared to simulate the odor associated with mixing of polymethacrylate , but the needle is not placed and cement is not injected.
  Interventions: Procedure: Sham procedure

INTERVENTIONS:
Device: percutaneous vertebroplasty — Using fluoroscopic guidance, the practitioner infiltrates the skin and subcutaneous tissues overlying the pedicle of the target vertebra or vertebrae with 1% lidocaine and infiltrates the periosteum of the pedicles with 0.25% bupivacaine (marcaine. For the vertebroplasty procedure, 11-gauge or 13-gauge needles are passed into the central aspect of the target vertebra or vertebrae. Bone cement is prepared on the bench and injected under constant fluoroscopy into the vertebral body. Injection is stopped when the PMMA reaches the posterior aspect of the vertebral body or leaks into an extraosseous space, such as the intervertebral disk or an epidural or paravertebral vein.
  Other Names: § 888.302713 Polymethylmethacrylate (PMMA) Bone Cement.
  Arms: percutaneous vertebroplasty
Procedure: Sham procedure — Using fluoroscopic guidance, the practitioner infiltrates the skin and subcutaneous tissues overlying the pedicle of the target vertebra or vertebrae with 1% lidocaine and infiltrates the periosteum of the pedicles with 0.25% bupivacaine (marcaine). During the sham intervention, verbal and physical cues, such as pressure on the patient's back, are given, and the methacrylate monomer (PMMA) is opened to simulate the odor associated with mixing of cement, but the needle is not placed and cement is not injected.
  Arms: Sham procedure

SUMMARY:
Background The standard care in patients with a painful osteoporotic vertebral compression fracture (VCF) is conservative therapy. Percutaneous vertebroplasty (PV), a minimally invasive technique, is a relatively new treatment option. Recent randomized controlled trials (RCT) provide conflicting results: two sham-controlled studies showed no benefit of PV while an unmasked but controlled RCT (VERTOS II) found effective pain relief at acceptable costs in patients with acute VCFs. A still ongoing masked RCT (VERTOS IV) focuses on acute VCFs defined as ≤ 6 weeks. VERTOS III focused on conservative treatment and found that half of patients still had disabling pain after 3 months or longer. These patients with sustained pain after 3 months may benefit from PV.

Objective To compare pain relief after PV with a sham intervention in selected patients with a chronic osteoporotic VCF ( three months or longer) using the same strict inclusion criteria as in VERTOS II an IV. Secondary outcome measures are back pain related disability and quality of life.

Methods The VERTOS V study is a prospective RCT with pain relief as primary endpoint. Inclusion criteria are a VCF of thoracic level 5 or lower with focal tenderness at fracture level, assessed by an internist on physical examination and a Visual Analogue Scale (VAS) score ≥ 5 for three months or longer, decreased bone density defined as T score ≤ -1 and age 50 years or older. 94 patients will be included, 47 in each arm. Crossovers are not allowed. Follow-up is at regular intervals during one year period with VAS score for pain as primary endpoint. Secondary endpoints are back pain related disability and quality of life measured with the Quality of Life Questionnaire of the European Foundation for Osteoporosis and physical function measured with the Roland Morris Disability questionnaire.

Conclusion Vertos V is a methodologically sound masked randomised sham controlled trial of vertebroplasty in patients with sustained pain 3 months or longer after a vertebral compression fracture.

ELIGIBILITY:
Inclusion Criteria:

* VCF on X-ray of the spine (minimal 15% loss of height)
* level of VCF Th5 or lower
* back pain ≥ 12 weeks at time of X-ray
* ≥ 50 years of age
* bone edema on MRI of the fractured vertebral body
* focal tenderness on VCF level
* decreased bone density T-scores ≤ -1

Exclusion Criteria:

* severe cardio-pulmonary condition
* untreatable coagulopathy
* systemic or local infection of the spine (osteomyelitis, spondylodiscitis)
* suspected alternative underlying disease (malignancy)
* radicular and/or cauda compression syndrome
* contra-indication for MRI

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-05; Primary Completion 2020-09-03 (Actual); Study Completion 2020-09-03 (Actual)

PRIMARY OUTCOMES:
Pain relief | 12 months
  Primary outcome will be pain score at 1 day, 1 week, and 1,3, 6 and 12 months after PV compared to baseline pain score. The questionnaire consist of the VAS score and questions about use of pain medication, pain location, and pain type. Other medical treatment and visits to alternative medical specialists, GP's and physical therapists are recorded and compared between groups. Patients are asked to fill out the VAS score and use of analgesics is recorded on a daily basis during the first month after randomization.

SECONDARY OUTCOMES:
Back pain related disability | 0, 1day, 1 week, 1,3,6,12 months
  Back pain related disability as measured with the Roland Morris Disability (RMD) Questionnaire. The Qualeffo is developed specifically for patients with osteoporosis. This questionnaire consists of 41 questions about: pain, physical function, social function, general health perception, and mental function. The RMD questionnaire is a disability questionnaire that measures the functional status of patients with back pain.
Quality of Life | 1 week, 1,3,6,12 months
  QOL as measured with the Questionnaire of the European Foundation for Osteoporosis (Qualeffo). The Qualeffo is developed specifically for patients with osteoporosis. This questionnaire consists of 41 questions about: pain, physical function, social function, general health perception, and mental function. The Qualeffo score ranges from 0 (best quality of life) to 100 (worst quality of life). This questionnaire will be completed at five measurement moments (before and at 1, 3, 6, and 12 months after the procedure).

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Carli, drs, Principal Investigator — Elisabeth Tweesteden Ziekenhuis/ SJG Weert; Paul Lohle, dr., Study Director — Elisabeth-TweeSteden Ziekenhuis
Locations (1):
- Elisabeth Tweesteden Ziekenhuis, Tilburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carli D, Venmans A, Lodder P, Donga E, van Oudheusden T, Boukrab I, Schoemaker K, Smeets A, Schonenberg C, Hirsch J, de Vries J, Lohle P. Vertebroplasty versus Active Control Intervention for Chronic Osteoporotic Vertebral Compression Fractures: The VERTOS V Randomized Controlled Trial. Radiology. 2023 Jul;308(1):e222535. doi: 10.1148/radiol.222535. PMID 37462495